CLINICAL TRIAL: NCT03754855
Title: Impact of Behavioral Factors on Treatment Adherence in a Sample of Rheumatoid Arthritis Patients
Acronym: MAINTAIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Association Aquitaine de Recherche Clinique en Rhumatologie (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/07
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; medication adherence; vaccination coverage; electronic health tools; diet
MeSH Terms: conditions — Arthritis, Rheumatoid; Medication Adherence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis patients: patients affected by RA according to ACR/EULAR 2010 criteria
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire

SUMMARY:
Rheumatoid arthritis (RA) care has been revolutionized in the last decade with the advent of biotherapies. Only 66% of treated patients are compliant. Nevertheless, studies analyzing the medication adherence in RA are rare. The aim of this study is thus to evaluate RA treatment adherence considering demographic data, vaccination coverage, feeding behavior and the use of e-health tools.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) care has been revolutionized in the last decade with the advent of biotherapies. The success of this therapeutic strategy is based on several factors, including the medication adherence. Whatever the method used, adherence evaluation is not sufficient, around 66% of the treated patients. Nevertheless, studies analysing the predictive factors of medication adherence in RA are rare.

RA patients are also educated about the infectious risk related to RA and treatments, and the importance of vaccination. These recommendations are not always respected by the patients, without knowing the exact factors leading to this decision. Furthermore, a lot of patients take personal initiatives without the agreement and the help of their practitioner, like diets or special feeding behaviors. Lastly, plenty of patients affected bv chronic diseases claim and use electronic health tools without any real evidence of the efficacy of such device.

The aim of this study is thus to evaluate RA treatment adherence considering demographic data, vaccination coverage, feeding behavior and the use of e-health tools.

ELIGIBILITY:
Inclusion Criteria:

* patient aged over 18 years old,
* affected by RA according to ACR/EULAR 2010 criteria,
* francophone,
* and informed about the aims of the study.

Exclusion Criteria:

* guardianship patient,
* patient who refuses to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged over 18 years old, affected by RA according to ACR/EULAR 2010 criteria
Sampling Method: Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who presented a good medication adherence according to the medication adherence questionnaire | At baseline (day 0)

SECONDARY OUTCOMES:
Proportion of patients vaccinated against influenza and pneumococcal bacteria | At baseline (day 0)
Proportion of reasons of non-vaccination, globally and for each type of vaccination. | At baseline (day 0)
Proportion of factors influencing rheumatologists to propose vaccination. | At baseline (day 0)
Proportion of vaccinated patients who present a good medication adherence to RA specific therapies | At baseline (day 0)
Proportion of patients using electronic health tools | At baseline (day 0)
Proportion of patients using electronic health tools who present a good medication adherence to RA specific therapies | At baseline (day 0)
Proportion of patients with a special diet, globally and by type of diet | At baseline (day 0)
Proportion of patients presenting functional bowel disorder | At baseline (day 0)
Proportion of patients with a special diet who present a good medication adherence to RA specific therapies | At baseline (day 0)
Number of patients with a good medication adherence, according to age | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to gender | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to socio-professional category | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to educational level | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to involvement in a patients association | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to alcohol and/or tobacco consumption | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to disease duration | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to rheumatoid factor and/or ACPA positivity | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to DAS28 score levels | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to actual RA treatments | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients with a good medication adherence, according to the use of alternative therapies (acupuncture and/or sophrology). | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires
Number of patients for each personality trait category | At baseline (day 0)
  Personality trait categories will be evaluated by the French version of Big Five Inventory questionnaire.
Number of patients with a good medication adherence, according to each personality trait category | At baseline (day 0)
  Medication adherence will be evaluated with medication adherence questionnaires. Personality trait categories will be evaluated by the French version of Big Five Inventory questionnaire.
Number of patients with a vaccination coverage, according to each personality trait category. | At baseline (day 0)
  Personality trait categories will be evaluated by the French version of Big Five Inventory questionnaire.
Number of patients with a special diet, according to each personality trait category | At baseline (day 0)
  Personality trait categories will be evaluated by the French version of Big Five Inventory questionnaire
Number of patients using electronic health tools, according to each personality trait category | At baseline (day 0)
  Personality trait categories will be evaluated by the French version of Big Five Inventory questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elise TRUCHETET, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - CHU de Bordeaux - service de rhumatologie, Bordeaux
  - Service de Rhumatologie, Clermont-Ferrand
  - Service de rhumatologie, Limoges
  - Service de rhumatologie, Montpellier
  - Service de Rhumatologie, Toulouse

IPD SHARING:
Plan to Share IPD: No